CLINICAL TRIAL: NCT05206565
Title: The Effect of Neurotization on Quality of Life and Sensory Restoration After Autologous Breast Reconstruction
Brief Title: Effect of Neurotization on QoL and Sensory Restoration
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Departmental hold on accrual, study never reopened and never accrued.
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021-0290; A539730 (Other: UW Madison); UW21028 (Other: UWCCC); Protocol Version 9/29/2021 (Other: UW Madison)
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Breast Reconstruction; Neurotization
Keywords: Quality of life

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Autologous with TRAM/DIEP flaps, with neurotization (Experimental): Autologous with TRAM/DIEP flaps, with neurotization
  Interventions: Procedure: Neurotization - Autologous Reconstruction with DIEP/TRAM
- Autologous with TRAM/DIEP flaps, without neurotization (No Intervention): Autologous with TRAM/DIEP flaps, without neurotization

INTERVENTIONS:
Procedure: Neurotization - Autologous Reconstruction with DIEP/TRAM — * Transverse Rectus Abdominis Muscle/Deep Inferior Epigastric Artery Flap Harvest - Prior to elevation of flaps in the suprafascial plane from using loupe magnification to identify medial and lateral row of perforators bilaterally, sensory nerves T10-12 are identified and dissected into the muscle bilaterally to prepare for nerve coaptation, nerves are divided at the level of the fascia where they are pure sensory nerves.
  * Chest Intercostal Nerve Harvest - During standard of care chest vessel dissection, intercostal nerves T3-4 are identified. After completion of vein coupling it will be determined whether neurotization can be performed or if autograft. Primary nerve coaptation will be performed if there is adequate length for direct end to end apposition.
  * Coaptation of nerve or nerve graft endings will be performed using 9-0 nylon suture in an interrupted fashion.
  Arms: Autologous with TRAM/DIEP flaps, with neurotization

SUMMARY:
This is a single-site, randomized, double-blinded trial to assess whether neurotization following autologous breast reconstruction in patients with breast cancer increases quality of life and sensation in the breast compared to breast reconstruction without neurotization. 50 participants will be enrolled and can expect to be on study for up to 18 months after reconstruction surgery.

DETAILED DESCRIPTION:
In 2019, nearly one third of cancers diagnosed in the United States were breast cancers. Per the Plastic Surgery procedural statistics from the American Society of Plastic Surgery database, that same year approximately 107,000 patients decided to pursue either alloplastic (ex. Tissue expander or implant based) or autologous (ex. Transverse Rectus Abdominis Muscle (TRAM), Deep Inferior Epigastric Perforator (DIEP) flaps) breast reconstruction, an increase of 5% from 2018. Over the past few decades, as surgical techniques have continued to improve, postoperative concerns have transitioned towards the patient's aesthetic outcome and satisfaction. While the appropriate size, shape, and symmetry of the breast are crucial goals to achieve, another issue facing patients is that without sensation the reconstructed breast does not feel like their own. In most patients there is diminished, if not absent, sensation in the reconstructed breast. The lack of sensation can not only put patients at risk of injury, but also can impact their lives sexually and socially.

The goal of this randomized, double-blinded study is to prospectively evaluate the impact of neurotization on breast-specific quality of life in patients who have undergone autologous reconstruction. Secondary objectives are to also look at additional health-related quality of life outcomes using validated surveys (e.g. PROMIS and NIH Toolbox). These NIH-funded surveys will be analyzed to assess factors important to surgical impact on physical function, mental function, social function, pain, and sexual function. Finally, investigators will objectively measure differences in sensation. Investigators hypothesize that breast neurotization will improve both breast- and health-related patient quality of life outcomes as well as objective sensation. The duration of this study is expected to be approximately 48 months in order to recruit an appropriate number of patients and have adequate postoperative follow up.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide informed consent
* The patient is ≥ 18 years
* Patients presenting to UW Health who have had or will have unilateral or bilateral mastectomy (therapeutic or prophylactic) and are planning to undergo autologous reconstruction with TRAM/DIEP will be included

Exclusion Criteria:

* Patient is non-English speaking
* Patient is known or believed to be pregnant
* Patient is a minor (individuals <18 years old)
* Patient is a prisoner
* Individuals unable to give consent due to another condition such as impaired decision-making capacity
* Autologous reconstruction where the flap is buried (e.g. there is no autologous skin exposed for sensation testing)
* Patient is a male
* Any patient with: diabetic neuropathy, thyroid disorders, collagen vascular disease, alcoholism, pernicious anemia, or any other severe underlying peripheral neuropathy
* Women with recurrent breast cancer
* Women who have undergone previous breast reconstructive procedures
* Not suitable for study participation due to other reasons at the discretion of the investigators
* Patient is currently lactating
* History of radiation therapy
* Patient undergoing a latissimus dorsi flap for reconstruction
* Patient undergoing alloplastic reconstruction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study population will consist of subjects with breast cancer who are scheduled for breast reconstruction and meet all inclusion/exclusion requirements.
Enrollment: 0 (Actual)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Breast-Q® score in participants who have undergone autologous reconstruction with TRAM/DIEP flaps with and without neurotization | approximately 12 months after reconstruction
  Self-reported, breast-specific health-related QoL(Quality of life) via use of the Breast-Q® in participant with breast cancer who have undergone autologous reconstruction with TRAM/DIEP flaps with and without neurotization.
  This score represents questionnaires about different domains and each question has four possible dimensions. The values of these dimensions varies from 1 to 4 (Likert Scale). The sum of each domain raw score scale will be plotted in the Breast Q Conversion Table to convert the summed domain score to a Equivalent Rasch Transformed Score with values ranging from 0 (worst) to 100 (best).

SECONDARY OUTCOMES:
Change in Breast-Q® score in participants who have undergone autologous reconstruction with TRAM/DIEP flaps with and without neurotization | Baseline(pre-operative), approximately 1-3 weeks, 6 weeks, 3 months, 6 months, 12 months, and 18 months after the reconstruction
  Self-reported, breast-specific health-related QoL(Quality of life) via use of the Breast-Q® in participant with breast cancer who have undergone autologous reconstruction with TRAM/DIEP flaps with and without neurotization.
  This score represents questionnaires about different domains and each question has four possible dimensions. The values of these dimensions varies from 1 to 4 (Likert Scale). The sum of each domain raw score scale will be plotted in the Breast Q Conversion Table to convert the summed domain score to a Equivalent Rasch Transformed Score with values ranging from 0 (worst) to 100 (best).
Change in Ability to Participate in Social Roles and Activities assessed by the PROMIS SF8a score in participants who have undergone autologous reconstruction with TRAM/DIEP flaps with and without neurotization | Baseline(pre-operative), approximately 1-3 weeks, 6 weeks, 3 months, 6 months, 12 months, and 18 months after the reconstruction
  The Patient-Reported Outcome Measurement Information System (PROMIS) Ability to Participate in Social Roles and Activities SF8a is a self-administered instrument to assess perceived ability to perform one's usual social roles and activities. Items are worded negatively in terms of perceived limitations, but responses are reverse-coded so that higher scores represent fewer limitations (better abilities). The item bank does not use a time frame (e.g. over the past seven days) when assessing ability to participate in social roles and activities.
Change in Pain Interference assessed by PROMIS SF8a score in participants who have undergone autologous reconstruction with TRAM/DIEP flaps with and without neurotization | Baseline(pre-operative), approximately 1-3 weeks, 6 weeks, 3 months, 6 months, 12 months, and 18 months after the reconstruction
  The Patient-Reported Outcome Measurement Information System (PROMIS) Pain Interference SF8a is a self-administered instrument that assesses the interference of pain on daily activities. Participants are asked to respond to questions regarding the extent of their pain. Responses range from 1 to 5, where 1 represents "not at all" and 5 represents "very much". A lower score indicates the least amount of pain interference.
Change in PROMIS Psychosocial Illness Impact-Positive SF8a score in participants who have undergone autologous reconstruction with TRAM/DIEP flaps with and without neurotization | Baseline(pre-operative), approximately 1-3 weeks, 6 weeks, 3 months, 6 months, 12 months, and 18 months after the reconstruction
  Measures the direct positive psychosocial effect related to illness using Computer Adaptive Testing (CAT) with higher scores reflecting better outcomes.
Change in PROMIS Psychosocial Illness Impact-Negative SF8a score in participants who have undergone autologous reconstruction with TRAM/DIEP flaps with and without neurotization | Baseline(pre-operative), approximately 1-3 weeks, 6 weeks, 3 months, 6 months, 12 months, and 18 months after the reconstruction
  Measures the direct negative psychosocial effect related to illness using Computer Adaptive Testing (CAT) with higher scores reflecting worse outcomes.
Change in Pressure-Specified Sensory Device (PSSD) score in participants who have undergone autologous reconstruction with TRAM/DIEP flaps with and without neurotization | Baseline(pre-operative), approximately 1-3 weeks, 6 weeks, 3 months, 6 months, 12 months, and 18 months after the reconstruction
  The PSSD Sensory Score is based on 1-point static and 2-point static pressure thresholds and 2- point distances. Cutaneous pressure thresholds and inter-prong distances are reported by the PSSD and determined to be normal or abnormal at a 99% confidence limit based on age (</= 45, or >45). These results correlate to a grading scheme which combines 1- and 2-point static pressure threshold with 2-point distance. An increase of greater than or equal to 1 grade from baseline as measured with the PSSD will be considered a meaningful change. The grading scale integrates normative data for each PSSD testing site.
Change in mean monofilament value in participants who have undergone autologous reconstruction with TRAM/DIEP flaps with and without neurotization | Baseline(pre-operative), approximately 1-3 weeks, 6 weeks, 3 months, 6 months, 12 months, and 18 months after the reconstruction
  Each monofilament value represents the logarithm of the force in milligrams required to bend the monofilament. Therefore, a thinner monofilament requires less pressure to bend and, if felt by the participant, represents improved one-point static discrimination compared to a participant who is not able to feel it.
  Perpendicular pressure will be applied to the same spot until monofilament bending is noted each time for a duration of 1.5 s, three times in succession, with intervals of 1.5 s. Testing will start with the thinnest monofilament and progress to monofilaments of increasing pressure until touch is identified in at least one out of three times by the participant. Participants will be asked to lay on their back and close their eyes, and measurements will take place in a quiet room. The different sites will be tested in a random sequence to ensure touch at a particular site cannot be predicted.
Change in number of touch sensitive breast locations in participants who have undergone autologous reconstruction with TRAM/DIEP flaps with and without neurotization | Baseline(pre-operative), approximately 1-3 weeks, 6 weeks, 3 months, 6 months, 12 months, and 18 months after the reconstruction
  The participant will be tested at 9 different spots on the breast and the number of locations on the breast participant are able to detect the filament will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Brett F Michelotti, MD, Principal Investigator — University of Wisconsin, Madison

IPD SHARING:
Plan to Share IPD: No